CLINICAL TRIAL: NCT00101140
Title: Phase II Study of Haploidentical Allogeneic Peripheral Blood Stem Cell Transplantation in Patients With High-Risk Acute Myeloid Leukemia in First Remission
Brief Title: Donor Stem Cell Transplant in Treating Patients With Acute Myeloid Leukemia in Remission
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000405838; ECOG-E1903
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Adult Acute Erythroid Leukemia; Adult Acute Monoblastic and Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia
Keywords: adult erythroleukemia (M6a); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myelomonocytic leukemia (M4)
MeSH Terms: conditions — Leukemia, Erythroblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Megakaryoblastic, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute | interventions — Antilymphocyte Serum; fludarabine phosphate; Thiotepa; Biological Therapy; Drug Therapy; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: anti-thymocyte globulin
Drug: fludarabine phosphate
Drug: thiotepa
Procedure: biological therapy
Procedure: bone marrow ablation with stem cell support
Procedure: chemotherapy
Procedure: non-specific immune-modulator therapy
Procedure: peripheral blood stem cell transplantation
Procedure: radiation therapy

SUMMARY:
RATIONALE: A peripheral stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy or radiation therapy. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving total-body irradiation together with fludarabine, thiotepa, and antithymocyte globulin before transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well a donor stem cell transplant works in treating patients with acute myeloid leukemia in remission.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and antileukemia activity of haploidentical allogeneic peripheral blood stem cell transplantation in patients with high-risk acute myeloid leukemia in first remission.

Secondary

* Determine the early treatment-related mortality (before day 100) of patients treated with this regimen.
* Determine the incidence of acute graft-versus-host disease in patients treated with this regimen.
* Determine the incidence of graft failure in patients treated with this regimen.
* Correlate a mismatch in the expression of the natural killer cell inhibitory receptors CD158a and CD158b with engraftment and disease recurrence in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive a preparative regimen comprising total-body irradiation twice on day -8; fludarabine IV over 30 minutes on days -7 to -3; thiotepa IV over 2 hours twice on day -7; and antithymocyte globulin IV over 4-6 hours on days -5 to -2. Patients undergo haploidentical allogeneic peripheral blood stem cell transplantation on day 0.

Patients are followed at day 100, at least monthly for 2 years, and then periodically for 3 years.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study within 2.2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed acute myeloid leukemia of 1 of the following subtypes:
* Acute myeloblastic leukemia (M0, M1, M2)
* Acute myelomonocytic leukemia (M4)
* Acute monocytic leukemia (M5)
* Acute erythroleukemia (M6)
* Acute megakaryocytic leukemia (M7)
* Must have 1 of the following karyotypic abnormalities at the time of diagnosis:
* Complex cytogenetic abnormalities (≥ 3 cytogenetic clones)
* Abnormalities of chromosome 5 [-5 or del(5q)]
* Abnormalities of the long (q) arm of chromosome 3, 9, 11, 20, or 21
* Abnormalities of the short (p) arm of chromosome 17, monosomy 7, t(9;22), or t(6;9) (8)
* In morphologic first complete remission*, as evidenced by all of the following for ≥ 4 weeks before study entry:
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Leukemic blasts not present in the peripheral blood
* Cellularity of bone marrow biopsy > 20% with maturation of all cell lines
* Less than 5% blasts by bone marrow biopsy
* No extramedullary leukemia, such as CNS or soft tissue involvement NOTE: *Reduced hemoglobin concentration or hematocrit has no bearing on remission status
* Haploidentical (3/6 or 4/6 antigen matched [A, B, and DR]) family donor available

PATIENT CHARACTERISTICS:

Age

* 18 to 59

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* AST < 2 times upper limit of normal

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* Ejection fraction > 40% by MUGA or echocardiogram
* None of the following within the past 3 months:
* Myocardial infarction
* Significant congestive heart failure
* Significant cardiac arrhythmia

Pulmonary

* FEV_1 and DLCO > 50% of predicted

Immunologic

* HIV negative
* No active or unresolved infection
* No evidence of invasive fungal infection (e.g., positive blood or deep tissue cultures or stains)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No organ damage
* No other medical problem that would preclude study participation
* No other currently active tumor that would likely interfere with study treatment or that would likely compromise the patient's morbidity or mortality

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent routine use of filgrastim (G-CSF) or sargramostim (GM-CSF) to accelerate hematopoietic recovery post-transplantation

Chemotherapy

* More than 4 weeks since prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Litzow, MD, Study Chair — Mayo Clinic; Jacob M. Rowe, MD — Rambam Health Care Campus